CLINICAL TRIAL: NCT05637008
Title: Determining Key Clinical Predictors for Chronic Ankle Instability and Return to Sports With Cost of Illness Analysis: a Prospective Cohort Study
Brief Title: Development of Chronic Ankle Instability After Acute Ankle Sprain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University of Ulster (Other); Bern University of Applied Sciences (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dirk Vissers, Professor, Universiteit Antwerpen
Other Study IDs: 1785
Record Dates: First submitted 2022-10-19; First posted 2022-12-05 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Ankle Sprains
Keywords: Ankle sprain; rehabilitation; sports injury; chronic ankle instability
MeSH Terms: conditions — Ankle Injuries; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational prospective cohort study is to determine key clinical predictors for chronic ankle instability and return to sports in patients who suffered an acute ankle sprain.

The researchers will evaluate clinical outcome measures and patient reported outcome measures on 3 test moments and at 12 months of follow-up.

DETAILED DESCRIPTION:
In this prospective cohort study, 4 different measurement time points will be used: 7-14 days, 6 weeks, 12 weeks and 12 months after the initial ankle sprain event. The researchers will include physically active people that engage in sports regularly, who recently suffered an acute ankle sprain. Recruitment will be done via hospital emergency departments, casualty departments and sports injury clinics, GP's, sports federations and social media.

The researchers will only use outcome measurements that are applicable in clinical practice, and patient reported outcome measures to evaluate the participants. The main outcome of this study is the development of chronic ankle instability, based on published criteria. The researchers aim to determine which clinically applicable outcome measures are key determinants for the development of chronic ankle instability. A secondary outcome is successful return to sports, with the objective to determine key clinically applicable determinants for successful recovery and return to sports.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Acute ankle sprain: <7 days
* Athletes (recreational or professional)
* Previous ankle sprain >12 months

Exclusion Criteria:

* Recurrent ankle sprain
* Ankle fracture
* Chronic ankle instability
* High ankle sprain (syndesmosis)
* A history of ankle or foot operations
* Other lower limb injuries and/or complaints
* Severe ocular impairments
* Any neurological, cardiac, vascular or metabolic disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We aim to recruit physically active participants - at least two organized sports sessions per week who sustained an acute ankle sprain.
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic ankle instability | 12 months
  Based on the predetermined criteria of the International Ankle Consortium, participants will have developed chronic ankle instability or not.
  https://www.jospt.org/doi/10.2519/jospt.2013.0303 - table 1

SECONDARY OUTCOMES:
Ability to return to sports | 12 months
  When participants are able to return to full participation at the same level prior to the injury, participants will have achieved successful return to sports. This outcome will be documented in a dichotomous manner: yes/no

OTHER OUTCOMES:
Muscle strength | 6 weeks and 12 weeks post injury
  Isometric muscle strength of the ankle and hip will be assessed
Ligament integrity | 7-14 days post injury
  Ankle sprain severity grade (grade 1: ligament fibre stretch; Grade 2: partial ligament tear; grade 3: complete ligament rupture) will be evaluated using a portable ultrasound, manual ligament stress testing, patient's perception of the ankle sprain severity, and bruising and palpation.
The amount of physical activity per day | 14 days, 6 weeks and 12 weeks post-injury
  The participants will wear an activity tracker to asses the amount of physical activity per day (hours)
The amount of sleep per night | 14 days, 6 weeks and 12 weeks post-injury
  Participants will wear an activity tracker to asses the amount of sleep per night in hours
Range of motion | Week 6 and 12 post injury
  Weight-bearing lunge test will be used to assess ankle dorsiflexion. A digital goniometer will be used to assess ankle dorsiflexion, plantar flexion, inversion, eversion
Ankle proprioception | Week 6 and 12 post injury
  A fixed handheld dynamometer (HHD) will be used to assess force sense as a measure of proprioception.
  To evaluate joint position sense as a measure proprioception, the slope-box test will be used.
Sensorimotor function: functional dynamic balance | Week 6 and 12 post injury
  Functional dynamic balance: y-balance test Participant will reach as far as possible in three directions - anterior, posterolateral, posteromedial. The reaching distance will be calculated in proportion to the lower limb length and be reported in percentage.
Sensorimotor function: static balance | Week 6 and 12 post injury
  static balance by single-leg stance: foot-lift test Participants will stand 30 seconds on one leg, with eyes closed. The amount of errors (deviations, foot lifts, ground touches from other foot) will be the outcome.
Sensorimotor function: dynamic balance | Week 6 and 12 post injury
  Single-leg dynamic balance: side-hop test Participants will hop 10 times sideways medially and laterally over a 30-cm distance as fast as possible. Time to perform the 10 hops back and forth is the outcome.
Performance: t-test | Week 6 and 12 post injury
  T-test for quickness: Participants will have to take place at an indicated starting line. On the signal, they will have to run forwards to the centre cone, sidestep 5 meters to the right cone, sidestep 10 meters to the far left cone and then sidestep back 5 meters to the centre cone. Conclusively, participants have to run backwards back to the starting line. This test is performed as quickly as possible.
Performance: drop landing | Week 6 and 12 post injury
  -single-leg drop landing: participant will perform a single-leg drop landing from a 30 cm box. The outcome is the ability to perform.
Performance: long jump | Week 6 and 12 post injury
  - Standing long jump: the participant will perform a single-leg long jump, as far as possible. The jump distance will be the outcome.
Performance: drop vertical jump | Week 6 and 12 post injury
  * Drop vertical jump: Participant will perform a drop off a 30 cm box, with a subsequent jump as high as possible. Outcomes of this test are jump height, stiffness, reactive strength index and contact time
  * T-test for quickness
Pain intensity and location | 7-14 days, 6 weeks and 12 weeks post injury
  Pain will be assessed using a numeric pain rating scale for pain severity from 0-10. 0 indicates no pain, 10 indicates unbearable pain. Additionally we will ask participants to show the location of their pain.
Perceived instability | 7-14 days, 6 weeks, 12 weeks and 12 months post injury
  Cumberland Ankle instability Tool: this assessment tool provides a scale up to 30 points. The higher the score, the worse the perceived instability of the participant.
Ankle-specific abilities | 7-14 days, 6 weeks, 12 weeks and 12 months post injury
  Foot and ankle ability measure - questionnaire: The short version of the Foot and Ankle ability measure (Quick-FAAM) will be used to evaluate region-specific functional abilities. This questionnaire contains twelve items scored across a 5-point Likert scale. High score indicates the inability to perform the evaluated task.
Illness perception | 7-14 days, 6 weeks, 12 weeks and 12 months post injury
  Illness perception questionnaire: The Illness perception questionnaire (IPQ) quantitatively evaluates the five components of illness representation: illness identity, cause, timeline, consequences and management on a 10-point Lickert scale. The higher the score (10), the worse the participant perceives the injury.
Fear avoidance | 7-14 days, 6 weeks, 12 weeks and 12 months post injury
  Fear avoidance believes pertinent to physical activities and work will be quantitatively evaluated by the fear avoidance beliefs questionnaire on a 7-point Lickert scale (0-6). 0 = disagrees with statement; 6= agrees with statement. There are 16 statements.
Fear | 7-14 days, 6 weeks, 12 weeks and 12 months post injury
  The 11-questions version of Tampa Scale for Kinesiophobia (TSK-11) will be utilized to assess pain-related fear of physical movement and activity. Participants have to provide their opinion regarding 11 statements: 1. totally disagree, 2. disagree for some part, 3. agree for some part, 4. totally agree.
Life quality | 7-14 days, 6 weeks, 12 weeks and 12 months post injury
  To assesses quality of life by addressing five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, the EQ-5D-5L questionnaire will be employed. Each domain is scored across a 5-point Likert scale: 0= no problems, 1= slight problems, 2= moderate problems, 3= severe problems and 4= extreme problems.
Cost of illness | 7-14 days, 6 weeks, 12 weeks and 12 months post injury
  Participants will be asked to share both direct and indirect costs related to the ankle sprain during the full course of the follow-up. Participants who incur a recurrent ankle sprain will be asked about both costs all over again.
Presence/ absence of a recurrent ankle sprain | Every month until 12 months follow-up
  We will ask patients whether they sustained a recurrent ankle sprain by short message service. The outcome is dichotomous: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Vissers, Prof., Principal Investigator — Universiteit Antwerpen
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagemans J, Taeymans J, Kuppens K, Baur H, Bleakley C, Vissers D. Determining key clinical predictors for chronic ankle instability and return to sports with cost of illness analysis: protocol of a prospective cohort study. BMJ Open. 2023 May 10;13(5):e069867. doi: 10.1136/bmjopen-2022-069867. PMID 37164478